CLINICAL TRIAL: NCT00675051
Title: Effect of Endothelin-1 Receptor Blockade on Circulating Endothelial Microparticles Levels in Patients With Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Yerem Yeghiazarians, Professor of Clinical Medicine, University of California, San Francisco
Other Study IDs: H47369-31390
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Hypertension
Keywords: To determine if there is a trans-pulmonary gradient in the levels of EMPs in patients with PH; To determine if the EMPs measured at the pulmonary capillary wedge position correlates even more strongly with the severity of PH than the circulating levels; To determine if PH therapy with ET-1 receptor blocker will modify EMPs levels
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pulmonary hypertension is a progressive and life threatening condition. It is characterized by severe remodeling of the pulmonary vessel wall, obstructive plexiform lesions, multi-focal thrombosis, and enhanced vasoconstriction. All of these characteristics contribute to increased pulmonary vascular resistance.

Circulating endothelial microparticles (EMPs) play an integral role in the pathogenesis and perpetuation of pulmonary hypertension. Levels of EMPs are considered a reliable biological parameter of endothelial injury.

We propose to assess the evolution of both circulating and pulmonary venous EMPs in patients with PH. Assessments will be made before and after initiation of Endothelin-1 (ET-1) Receptor blocker therapy, and correlated to their patterns with the changes in mean PAP, the 6 Minutes Walking Distance test, and circulating Endothelin-1 values. Measurements of the endothelial microparticle circulating levels (assessed by flow cytometry methods) will be made before, 1 month and 3 months after initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient's + 18 years with suspected pre-capillary pulmonary hypertension
* Prescribed Endothelial - 1 receptor blocker

Exclusion Criteria:

* Currently taking endothelium-active vasodilator therapy.
* Hemoglobin and / or hematocrit level blood the lower normal limit.
* Left ventricle dysfunction (LVEF <50%)
* LV end-diastolic pressure > 15 mmHg)
* Recent history (<3 months) of pulmonary embolism
* Liver failure or abnormal liver function tests; aortic or mitral regurgitation or stenosis
* Current medication with endothelin-1 receptor antagonist, prostacyclin analogues or type 5 phosphodiesterase inhibitors.
* Subjects with conditions known to be associated with an increase in circulating endothelial microparticle numers, such as chronic renal failure (Creatinine Clearance < 50 ml/min/m2) acute coronary syndromes and uncontrolled system hypertension.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Precapillary Pulmonary Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, California, United States